CLINICAL TRIAL: NCT03575663
Title: Bronchial Challenge Testing in Asthma: The Effect of Mannitol Dry Powder Inhalation on Volatile Organic Compounds in Exhaled Breath
Brief Title: The Asthma Bronchial Challenge Study
Acronym: ABC
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Collaborators: University of Manchester (Other); Asthma UK Centre for Applied Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2229225
Record Dates: First submitted 2018-06-11; First posted 2018-07-02 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2018-04

CONDITIONS: Asthma
Keywords: Breathomics; Metabolomics; Exhaled breath test; Biomarker
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Volatile organic compounds obtained through sampling exhaled breath
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Indirect bronchial challenge — Mannitol dry powder inhalation
  Other Names: Osmohale / Aridol
Other: Sham bronchial challenge — Mock dry powder inhalation

SUMMARY:
This is a randomised, controlled, cross-over study to determine the effect of indirect bronchial challenge testing upon volatile organic compounds (VOCs) in the exhaled breath of adults with well-controlled, mild-to-moderate asthma.

Participants will undergo baseline evaluation including clinical history, spirometry, exhaled nitric oxide measurement (FeNO), phlebotomy (blood eosinophil count), and sampling of exhaled breath VOCs. Participants will be randomised to receive either an indirect bronchial challenge test using mannitol dry powder (MDP) or a sham bronchial challenge, followed by further sampling of breath VOCs. The study will consist of a consent visit and two assessment visits with participants allocated to receive one of the two challenges (MDP or sham) at each assessment. Data will be analysed to determine the effect of bronchial challenge upon exhaled breath VOC profiles.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18 or over
* Able to provide informed consent
* Self-report of asthma diagnosis from health professional
* Diagnostic confirmation meeting British Thoracic Society guidelines will be sought from primary care
* Non-smokers; or ex-smokers of at least two years duration with less than a ten pack year history
* Asthma Control Questionnaire score < 1.0
* Asthma treated according to level-1 to level-2 of British Thoracic Society treatment guidelines

Exclusion Criteria:

* Respiratory tract infection, asthma exacerbation or change in treatment step within the previous four weeks
* Major chronic cardiorespiratory disease other than asthma
* Significant comorbid condition
* Condition that may be compromised by repeated spirometry manoeuvres or induced bronchospasm
* Asthma Control Questionnaire score >1.0
* Asthma treated at level 3 of the treatment guidelines or higher
* Pregnant or nursing mothers
* Current smokers or 'vapers'
* Ex-smokers of < 2 years duration or > 10 pack years.
* Participating in a clinical trial of an investigational medicinal product (CTIMP).
* Unable to speak English.
* Low baseline lung function (FEV1 <1.50 litres or < 70% predicted value)
* Known hypersensitivity to mannitol, gelatin or strong anaphylactic response in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with well-controlled, mild asthma, managed in primary care and treated at level 1 to 2 of the British Thoracic Society treatment guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in exhaled breath profile | Immediately post-bronchial challenge
  Exhaled volatile organic compounds (VOCs) will be captured on sorbent material and analysed by gas chromatography-mass spectrometry. Post-bronchial challenge samples will be compared with baseline, pre-challenge samples. Differences in exhaled VOC profile will be assessed for significance.

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Peel, BSc, Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No